CLINICAL TRIAL: NCT02831972
Title: An Open-Label, 2-Period, Fixed Sequence Study to Determine the Effect of Multiple Oral Doses of Itraconazole on the Single Dose Pharmacokinetics of AG 120 in Healthy Adult Subjects
Brief Title: Drug-Drug Interaction Study of AG120 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG120-C-007
Record Dates: First submitted 2016-06-09; First posted 2016-07-13 (Estimated); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — ivosidenib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Period 1 (Experimental): A single oral dose of AG-120 will be administered at Hour 0 followed by PK sampling for 504 hours (21 days).
  Interventions: Drug: AG120
- Period 2 (Experimental): In Period 2, multiple oral doses of itraconazole will be administered once daily (QD) for 18 consecutive days (Days -4 to 14) with a single oral dose of AG-120 coadministered at Hour 0 on Day 1. PK sampling for AG-120 will be taken for 504 hours (21 days) following AG-120 dosing on Day 1. PK sampling will also be collected for itraconazole and its metabolite, hydroxy-itraconazole, from Day -2 up to Day 13.
  Interventions: Drug: AG120; Drug: Itraconazole

INTERVENTIONS:
Drug: AG120
Drug: Itraconazole
  Arms: Period 2

SUMMARY:
An Open-Label, 2-Period, Fixed Sequence Study to Determine the Effect of Multiple Oral Doses of Itraconazole on the Single Dose Pharmacokinetics of AG 120 in Healthy Adult Subjects. Period 1 consists of a single oral dose of AG-120 will be administered at Hour 0 followed by PK sampling for 504 hours (21 days). In Period 2, multiple oral doses of itraconazole will be administered once daily (QD) for 18 consecutive days with a single oral dose of AG-120 coadministered at Hour 0 on Day 1. PK sampling for AG-120 will be taken for 504 hours (21 days) following AG-120 dosing on Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, adult, male or female, 18 - 55 years of age, inclusive, at screening.
2. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose and throughout the study.
3. BMI ≥ 18.5 and ≤ 32.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. For a female of childbearing potential: either be sexually inactive (abstinent) for 14 days prior to the first dose and throughout the study or be using one of the following acceptable birth control methods:

   * non-hormone releasing intrauterine device for at least 3 months prior to the first dose and with either a physical (e.g. condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study.
   * surgical sterilization of the partner (vasectomy for 4 months minimum the first dose/dosing) and with either a physical (e.g. condom, diaphragm, or other) or a chemical (e.g., spermicide) barrier method from the time of screening and throughout the study.
   * two physical barrier method (e.g. condom, diaphragm, or other) with spermicide for at least 14 days prior to the first dose and throughout the study.

   In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 90 days following the last dose.
6. For a female of non childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to the first dose:

   * hysteroscopic sterilization;
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy. or be postmenopausal with amenorrhea for at least 1 year prior to the first dose and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status as per PI or designee judgment.
7. A non vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days beyond the last dose of study drug. (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to first dose of study drug. A male who has been vasectomized less than 4 months prior to study first dose must follow the same restrictions as a non vasectomized male).
8. If male, must agree not to donate sperm from the first dose until 90 days after the last dose.
9. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

1. Subject is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
6. History or presence of ventricular dysfunction or risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, family history of Long QT Syndrome).
7. Female subjects with a positive pregnancy test or lactating.
8. Positive urine drug or alcohol results at screening or each check in.
9. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
10. QTcF interval is >450 msec (males) or >460 msec (females) or has ECG findings deemed abnormal with clinical significance by the PI or designee at screening.
11. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non prescription medications, herbal remedies, or vitamin supplements beginning 14 days prior to the first dose and throughout the study. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study.
    * Any drugs known to be significant inducers of CYP enzymes and/or P gp, including St. John's Wort, for 28 days prior to the first dose and throughout the study. Appropriate sources will be consulted by the PI or designee to confirm lack of PK/pharmacodynamic interaction with study drug(s).
12. Has been on a diet incompatible with the on study diet, in the opinion of the PI or designee, within the 28 days prior to the first dose and throughout the study.
13. Donation of blood or significant blood loss within 56 days prior to the first dose.
14. Plasma donation within 7 days prior to the first dose.
15. Participation in another clinical study within 28 days prior to the first dose. The 28 day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
AG120 Area Under the Curve [AUC] | Period 2: itraconazole administered once daily (QD) for 18 consecutive days (Days -4 to 14) with a single oral dose of AG-120 coadministered at Hour 0 on Day 1. PK sampling for AG-120 will be taken for 504 hours (21 days)
AG120 Maximum Plasma Concentration [Cmax] | Period 2: itraconazole administered once daily (QD) for 18 consecutive days (Days -4 to 14) with a single oral dose of AG-120 coadministered at Hour 0 on Day 1. PK sampling for AG-120 will be taken for 504 hours (21 days)
Itraconazole Area Under the Curve [AUC] | Period 2: itraconazole administered once daily (QD) for 18 consecutive days (Days -4 to 14) with a single oral dose of AG-120 coadministered at Hour 0 on Day 1. PK sampling for AG-120 will be taken for 504 hours (21 days)
Itraconazole Maximum Plasma Concentration [CMAX] | Period 2: itraconazole administered once daily (QD) for 18 consecutive days (Days -4 to 14) with a single oral dose of AG-120 coadministered at Hour 0 on Day 1. PK sampling for AG-120 will be taken for 504 hours (21 days)

SECONDARY OUTCOMES:
Hydroxy-itraconazole Area Under the Curve [AUC] | Period 2: Day -2 up to Day 13
Hydroxy-itraconazole Maximum Plasma Concentration [CMAX] | Period 2: Day -2 up to Day 13

CONTACTS AND LOCATIONS:
Locations (1):
- Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No